CLINICAL TRIAL: NCT00162227
Title: US Sustiva Oral Liquid Expanded Access Program: an Open-label, Multicenter Expanded Access Study of the Liquid Formulation of Sustiva (Efavirenz, DMP 266)
Brief Title: An Expanded Access Study of Oral Liquid Efavirenz in the Treatment of Children With HIV Infection
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI266-913
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — efavirenz

INTERVENTIONS:
Drug: Efavirenz — Oral Solution, Oral 200 - 600 mg (weight based), once daily. Until further treatment with Sustiva Oral Solution is not warranted.
  Other Names: Sustiva; BMS-561525

SUMMARY:
This study is being conducted to assess the safety and tolerability of an oral liquid solution of Sustiva for antiretroviral therapy-naive or therapy-experienced HIV-1 infected children between the ages 3-16 who are failing or intolerant of current antiretroviral regimen and who are unable to swallow Sustiva capsules.

ELIGIBILITY:
Inclusion Criteria:

* Children 3-16 years of age
* Anti-retroviral naive or experienced
* Failing or intolerant to current Anti-retroviral regimen
* Limited available viable therapeutic options
* Inability to take capsules/tablets

Exclusion Criteria:

* Less than 10kg
* Failure on or concomitant use of other NNRTIs
* An active AIDS-defining opportunistic infection or disease
* More than two episodes of moderate to severe diarrhea or vomiting lasting more than four days within the past three months

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2000-09; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (29):
- United States (27):
  - Local Institution, Phoenix, Arizona
  - Lac & Usc Medical Center, Los Angeles, California
  - Local Institution, Washington D.C., District of Columbia
  - Children'S Diagnostic Treatment Center, Fort Lauderdale, Florida
  - Arnold Palmer Hospital For Children And Woman, Orlando, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - The Children'S Memorial Hospital, Chicago, Illinois
  - University Of Chicago, Chicago, Illinois
  - Lsu Health Sciences Center, New Orleans, Louisiana
  - Children'S Hospital, Boston, Massachusetts
  - University Of Massachusetts Medical School, Worcester, Massachusetts
  - The Wellness Center, Las Vegas, Nevada
  - Umdnj - New Jersey Medical School, Newark, New Jersey
  - Schneider'S Childrens Hospital, New Hyde Park, New York
  - Office Of John Montana, New York, New York
  - St Luke'S-Roosevelt Hospital Center, New York, New York
  - Women And Childrens Care Center, New York, New York
  - Harlem Hospital Center, New York, New York
  - State University Of New York At Stony Brook, Stony Brook, New York
  - Suny Upstate Medical University, Syracuse, New York
  - Bronx Municipal Hospital Center, The Bronx, New York
  - Montefiore Medical Center/Aecom, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Metro Health Medical Center, Cleveland, Ohio
  - Local Institution, Youngstown, Ohio
  - St Jude Children'S Research Hospital, Memphis, Tennessee
  - Local Institution, Houston, Texas
- Puerto Rico (2):
  - Local Institution, Arecibo
  - Local Institution, San Juan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx